CLINICAL TRIAL: NCT01982110
Title: A Mindfulness Based Application for Smoking Cessation
Acronym: MBSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jennifer Kim Penberthy, Department of Psychiatry and Neurobehavioral Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17004
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Nicotine Dependence
Keywords: smoking cessation; mindfulness; behavioral intervention
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Therapy (Experimental): Craving to Quit mobile application is provided for participants
  Interventions: Behavioral: Mindfulness based smoking cessation
- Behavioral Smoking Cessation (Active Comparator): NCI Quit Pal via a mobile phone application is provided for participants
  Interventions: Behavioral: Behavioral Smoking Cessation intervention

INTERVENTIONS:
Behavioral: Mindfulness based smoking cessation — Mindfulness based interventions are provided via a mobile phone application.
  Other Names: Craving to Quit
  Arms: Mindfulness Based Therapy
Behavioral: Behavioral Smoking Cessation intervention — Behavioral Smoking Cessation intervention is a behaviorally based intervention is provided via a mobile phone application.
  Other Names: Behavioral therapy; Cognitive Behavioral therapy; NCI QuitPal
  Arms: Behavioral Smoking Cessation

SUMMARY:
Cigarette smoking is the leading cause of preventable death and disability in the world. Although over 70% of smokers want to quit, fewer than 5% achieve this goal annually. Additional effective, safe, and accessible treatments for nicotine dependence are needed due to the low abstinence rates (20-30%) achieved in behavioral therapies, the unappealing side effects of pharmacotherapy, and the frequent lack of accessibility to treatment. Recent evidence supports the central role of craving in maintaining nicotine dependence, and neither behavioral nor replacement therapies directly target the relationship between cravings and smoking. Mindfulness therapy has been found to be effective in teaching strategies to decouple the association between craving and smoking. Mindfulness based smoking therapy (MT) has preliminary support for reducing consumption in smokers, and Dr. Judson Brewer has recently translated this program into a mobile device application (app) for smoking cessation. With Dr. Brewer's consultation, we propose to assess the feasibility of implementation of a MT mobile application in local hospital and community clinics and the effectiveness of the MT mobile application compared to a National Cancer Institute (NCI) QuitPal behavioral change group. We will examine smoking results at end of treatment and 2 and 6 month follow-up as well as the role of craving. If MT smoking cessation is determined to be effective in a mobile phone application, this finding will be a significant step in providing an additional effective and safe treatment for smokers wishing to quit or cut down on their intake, and will be especially important in providing treatment options for marginalized or hard-to-access individuals wishing to reduce cigarette intake.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of preventable death and disability in the world, accounting for 10% of all deaths. In the US, smoking costs more than $193 billion in health care costs and lost productivity per year. Although over 70% of smokers want to quit, fewer than 5% achieve this goal annually. Mainstay behavioral treatments for smoking have focused on teaching individuals to avoid cues, foster positive affective states, develop lifestyle changes that reduce stress, divert attention from cravings, substitute other activities for smoking, learn cognitive strategies that reduce negative mood and develop social support mechanisms. These have shown modest success, with abstinence rates between only 20-30% over the past thirty years. This is presumably due to the complex nature of the acquisition and maintenance of nicotine addiction, including associative learning mechanisms as well as positive and negative reinforcement. Over time, cues that are judged to be positive or negative can induce affective states, which can then trigger a craving to smoke. Though the centrality of craving remains controversial, evidence suggests that craving is strongly associated with smoking, which, mainly through the physiological properties of nicotine, results in the maintenance or improvement of positive or reduction of negative affective states. This sets up reinforcement loops by reinforcing memories between affect and smoking. Thus, attention has been focused on additional strategies to help people tolerate negative affect and cravings rather than avoiding cues or substituting activities, and recent research suggest that MT may decouple the association between craving and smoking, thus facilitating smoking cessation.

Mindfulness training (MT) targets affective or craving states by teaching individuals to observe aversive body and mind states instead of reacting to them with habitual reactions, thus allowing more adaptive, healthier responses. Mindfulness training (MT) has shown promise in reducing anxiety and depression and has recently been explored in the treatment of addictions. In a 2011 randomized controlled trial by Brewer, et al., individuals who received an 8- session MT vs. the American Lung Association's 8 session freedom from smoking (FFS) treatment, showed significantly greater rate of reduction in cigarette use and greater point prevalence abstinence rates during treatment and maintained these gains during follow up. FFS is a behavior modification program and includes stress reduction and relapse prevention. Although both treatment groups were assigned home practice as part of their treatment, only those who received mindfulness training demonstrated a significant association between home practice and smoking outcomes, suggesting that there was a specific benefit to mindfulness practice and that positive treatment outcomes for those in this group are not merely a result of greater enthusiasm or interest in quitting. The ability of MT to attenuate the relationship between craving and substance use has been observed in other studies as well. Elwafi, et al. (2012) demonstrated that people who practiced mindfulness more smoked less, regardless of their level of craving. Practicing mindfulness appears critical to MT treatment outcomes. These results suggest that MT may help individuals develop a tolerance to craving itself, thus over time acting to dismantle the addictive loop. To date, research in this area has been conducted in randomized clinical trials in structured laboratory settings only. Important next steps are to examine the effectiveness of MT treatments for smoking cessation in naturalistic environments and to utilize methods of delivering treatment in real world settings that will facilitate compliance with mindfulness practice and thus improve treatment outcomes - for example, via a mobile device application. Additionally, trials comparing MT to alternative treatment approaches typically offered in outpatient clinics such as support groups, acupuncture, individual counseling, or nicotine replacement therapies are lacking. Mindfulness based (MT) smoking cessation has been adapted to a mobile device application called "Craving to Quit" based on the work done by Brewer and will be the mindfulness intervention used in this study. Standardization and implementation via a mobile application is a logical and necessary next step in the dissemination of treatment and will potentially provide access to an effective smoking cessation program for persons who may not otherwise be able to access treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* 18 years of age or older
* Smoke an average of a minimum of five cigarettes per day
* Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of mindfulness techniques
* Express a wish to quit smoking
* A score at least in the "contemplation" range, as assessed via the Readiness to Change questionnaire (Heather & McCambridge, 2013)
* Willingness to participate in mindfulness techniques
* Able to attend all clinic visits without interruption

Exclusion Criteria:

* Any current Axis I DSM-IV-TR psychiatric disorder other than alcohol abuse, marijuana abuse, or nicotine dependence that, in the clinician's opinion, warrants treatment or would preclude safe participation in the protocol, including, but not limited to: psychosis, schizophrenia, dementia, schizotypal personality disorder, borderline personality disorder, bipolar disorder, primary diagnosis of eating disorder, or chronic suicidality or homicidality
* Serious medical comorbidity requiring medical intervention or close supervision, including seizures, pacemakers, heart transplant, severe arrhythmias, or active atrial fibrillation
* Suicide attempt in the last thirty days
* Gross neurological disease
* Mental retardation, which will be assessed by the PI, postdoctoral fellows, and doctoral students in clinical psychology
* Minors below the legal smoking age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Smoking behavior | 6 months
  We will assess number of cigarettes smoked and CO levels

SECONDARY OUTCOMES:
Craving | 6 months
  We will assess levels of craving to smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Penberthy, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700